CLINICAL TRIAL: NCT03330119
Title: Determining the Effect of an "Alternate Recovery Protocol" Versus Current Standard of Care After Cesarean Section
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of Funding/ Resident in charge graduated
Sponsor: Brest, Norman A., M.D. (Other)
Responsible Party: Principal Investigator, Norman A. Brest, Principle Investigator, Brest, Norman A., M.D.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: F/N-R17-3732L
Record Dates: First submitted 2017-10-24; First posted 2017-11-06 (Actual); Results first posted 2021-03-02 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-03

CONDITIONS: Pregnancy Related; Narcotic Use
Keywords: Pregnancy; cesarean section; enhanced recovery; narcotic use
MeSH Terms: interventions — Enhanced Recovery After Surgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Alternate Management (Experimental)
  Interventions: Drug: Alternate Management
- Control (Placebo Comparator): The regular Lankenau cesarean section order set.
  Interventions: Drug: Control

INTERVENTIONS:
Drug: Alternate Management — With the alternate management protocol, the pre-operative order set is the same, with the addition of a single preoperative dose of acetaminophen 1 g IV x1, gabapentin 600 mg PO x1, and ondansetron 8 mg IV x1. Post-operatively, patients receive the same ketorolac 30mg x 9 doses every 6 hours, as well as acetaminophen 975 mg every 6 hours, both given standing. These two are timed so the patient is receiving one of the two medications every 3 hours during their inpatient stay. After 9 doses of ketorolac, the patient receives 600mg of ibuprofen PO, also given standing, instead of the ketorolac. If the patient requires narcotics, they may receive them on an as needed basis. IV fluids are running at 80 cc/ hour. Patients are encouraged to ambulate, including the evening of the surgery, have their foley catheter removed 12 hours post-operatively, and can have a regular diet immediately.
  Other Names: Enhanced Recovery
  Arms: Alternate Management
Drug: Control — The regular Lankenau cesarean section order set includes routine vital signs, labs, IV fluids, and fetal heart monitoring. Post standard cesarean section orders include IV fluids running at 125 cc/ hour, along with routine post-partum care. In terms of pain control, most patients receive 9 doses of 30mg of IV ketorolac every 6 hours, along with hydromorphone, oxycodone/acetaminophen, or a hydromorphone PCA, per patient or attending request.
  Arms: Control

SUMMARY:
This randomized controlled trial will compare two different approaches to patient recovery after cesarean section: the current standard of care versus an alternate management protocol. The goal of this study is to investigate whether an "alternate management" protocol after cesarean sections will yield the same results as alternate management in other surgical fields, including decreased narcotic consumption and quicker return of bowel function, without compromising patient morbidity or satisfaction.

The investigators will assess postoperative narcotic consumption as the primary outcome. Secondary outcomes will be return of bowel function, length of hospital stay, pain control, patient satisfaction, post-operative complications, and overall morbidity and mortality.

Hypothesis: Initiating the alternate management protocol for cesarean sections will decrease narcotic consumption and hasten return of bowel function, without compromising patient satisfaction, level of pain control, or post-operative morbidity.

DETAILED DESCRIPTION:
"Enhanced recovery" is a multi-modal, evidence based approach to peri-operative care, with the goal of accelerating recovery and return to normal activity after surgery. Initially introduced in colorectal surgery, some of the key changes in management include: preoperative patient education, reduction in preoperative fasting, peri-operative euvolemia, early removal of urinary catheters, multimodal and standing analgesia, early postoperative mobilization, and earlier return to a regular diet. Results have shown stable pain control with a decrease in narcotic consumption, a quicker return of bowel function, and decreased length of hospital stay and cost with no change in level of patient satisfaction, morbidity, or readmission rate. The thought is that these interventions speed recuperation by attenuating the stress response associated with surgery, subsequently decreasing time spent in the hospital and improving quality of life.

The largest retrospective cohort study demonstrating the successful implementation of the "enhanced recovery" protocol in gynecology was conducted at the Mayo Clinic, published in 2013. This protocol was created by general gynecologists, gynecology oncologists, urogynecologists, anesthesiologists, pharmacists, and nursing, and was initiated as a quality improvement project. This "enhanced recovery" protocol was used as the template for our alternate management order set. The results showed an 80% reduction in opioid consumption, stable pain scores and patient satisfaction, a 1 day earlier return of bowel function, and 4 day reduction in hospital stay with subsequent significant cost savings. An obstetric alternate management protocol was created at Lankenau, trying to incorporate the most current recommendations in "enhanced recovery" while accounting for issues unique to obstetric patients. This protocol is currently being used by certain obstetricians.

The only literature published on "enhanced recovery" being implemented in the field of obstetrics was an observational study conducted with 708 C-sections at the Jessop Wing Obstetric Unit, in Sheffield, England, published in 2015. See below for the protocol used. The development of an obstetric "enhanced recovery" plan resulted from a desire for earlier discharge following cesarean section, due to pressure on national health service budgets to cut costs. There was an increase in day 1 discharges following uncomplicated cesarean sections from 1.6% to 25 % with the above mentioned protocol, and a stable 30 day readmission rate. Their conclusion was that "an enhanced recovery program was successfully implemented… Many of the interventions were straightforward and could be adopted easily elsewhere."

A somewhat controversial element of the "enhanced recovery" protocol is the use of gabapentin in pregnancy. Gabapentin is a Category C drug, meaning that risk cannot be ruled out in pregnancy and that the drug should be given if potential benefits outweigh potential risks. Our alternate management order set includes giving 1 dose of 600mg of pre-operative gabapentin. There have been many papers documenting its safety when given as a single dose pre-operatively. A randomized controlled trial published in 2011 in the Society of Obstetric Anesthesia and Perinatology, evaluated the peri-operative use of gabapentin for cesarean sections. Neonatal outcomes were evaluated for the gabapentin group, involving 600mg pre-operatively, as well as the placebo group. There was no significant difference in neonatal outcomes. A second study published in 2015 in the American Society of Anesthesiologists also showed no difference in neonatal outcomes with a single pre-operative dose of 600mg gabapentin. Lactmed, a database that lists drugs and dietary supplements that may affect breastfeeding, endorsed by the American Academy of Pediatrics, states that "maternal doses of gabapentin up to 2.1 grams daily produce relatively low levels in infant serum," and that " a single PO dose of 600 mg prior to cesarean section appeared to have no effect on breastfeeding initiation."

Given that the national cesarean section rate in the United States is 32.2%, implementing an "enhanced recovery" protocol in obstetrics could have a huge impact on care for women in the post-partum period. The widespread adoption of "enhanced recovery" stems from evidence showing reduced narcotic consumption, earlier return to normal activities, and even reduced morbidity in some studies. From a post-partum standpoint, given the increased risk of DVT until 6 weeks post-partum, and the additional increased risk after cesarean section, encouraging ambulation and return to normal activity seems beneficial. Also, the potential to decrease narcotic use has great implications in both the post- partum and post- operative period. The CDC has recently published guidelines on prescribing opioids, given that opioid abuse is a growing epidemic in this country. The American Congress of Obstetricians and Gynecologist had responded saying that physicians would try to combat the use of prescription opioids across the country and that they should be using current best prescribing practices and all possible options for multimodal pain relief. Additionally, the American Academy of Pediatrics published an update to their Transfer of Drugs and Therapeutics in Human Breast Milk Series in 2013. The AAP states that acetaminophen and ibuprofen should be used as first line therapy for post-partum pain management, and discourages the use of codeine, hydrocodone, and oxycodone when breast feeding. One study found that as high as 20% of infants exposed to oxycodone through breast milk had central nervous system depression. Also, the state of Pennsylvania has started a breast feeding quality improvement project, called the Keystone 10 Initiative, developed by the department of health. The goal is to promote and support breastfeeding to "improve the health of mothers and babies," through changes such as more skin to skin contact and less time infants spend in the nursery. Given that the most common side effect of narcotic use is somnolence, seen up to 42% of the time, this may interfere with the mother's ability to care for her newborn. Therefore, it is clear that an "enhanced recovery" protocol after cesarean sections has potential to improve care post-operatively and post-partum on multiple levels.

Methods:

A randomized control pilot study will be performed with the primary outcome of narcotic utilization in the post-operative period. After IRB approval, patients will be recruited for the study in the outpatient setting or upon their arrival to the labor and delivery floor, for their scheduled cesarean section. They will be consented by the principal investigator, or his designee. Consent for the study will include a series of questions related to the exclusion criteria listed below in addition to the risks and benefits of the study. The patient will be randomized to either the alternate management group, or the standard cesarean section group, via computer randomization.

The regular Lankenau cesarean section order set includes routine vital signs, labs, IV fluids, and fetal heart monitoring. Post standard cesarean section orders include IV fluids running at 125 cc/ hour, along with routine post-partum care. In terms of pain control, most patients receive 9 doses of 30mg of IV ketorolac every 6 hours, along with hydromorphone, oxycodone/acetaminophen, or a hydromorphone PCA, per patient or attending request.

With the alternate management protocol, the pre-operative order set is the same, with the addition of a single preoperative dose of acetaminophen 1 g IV x1, gabapentin 600 mg PO x1, and ondansetron 8 mg IV x1. Post-operatively, patients receive the same ketorolac 30mg x 9 doses every 6 hours, as well as acetaminophen 975 mg every 6 hours, both given standing. These two are timed so the patient is receiving one of the two medications every 3 hours during their inpatient stay. After 9 doses of ketorolac, the patient receives 600mg of ibuprofen PO, also given standing, instead of the ketorolac. If the patient requires narcotics, they may receive them on an as needed basis. IV fluids are running at 80 cc/ hour. Patients are encouraged to ambulate, including the evening of the surgery, have their foley catheter removed 12 hours post-operatively, and can have a regular diet immediately.

The morphine equivalent score will be used to calculate total narcotic use while the patient remains as an inpatient. Secondary outcomes will include presence of flatus, assessed at 8 hour intervals, and pain via the visual analogue scale. Patient satisfaction will be assessed using the validated survey used in the Mayo Clinic Trial, to be filled out prior to discharge. Post-operative complications and readmissions will be noted during the inpatient stay. Information regarding patient satisfaction, pain score, and presence of flatus will be gathered by nursing, and will be self-reported by the patient. Total narcotic use will be calculated.

Sample Size: 65 standard recovery patients, 65 alternate management patients Using the Vanderbilt power calculator, and an alpha value of 0.5, and a beta of 20%, to achieve a 50% reduction in narcotic use, approximately 65 patients will be required in each group. The investigators will perform an interim analysis on our data, after 65 subjects have been recruited, both for efficacy and assessment of any adverse outcomes. This will help the investigators determine fewer or more patients are needed in order to achieve a statistically significant difference in narcotic consumption.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo a cesarean section

Exclusion Criteria:

* Existing diagnosis of chronic pain
* Need to undergo a vertical skin incision
* AST > 50; ALT > 70
* Platelets below 80,000 on admission
* Need to undergo general anesthesia
* Tubal ligation at time of Cesarean section
* Prior or known allergy to any of the medications being utilized in this study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1494 (Actual)
Dates: Start 2017-10-04 (Actual); Primary Completion 2018-06-20 (Actual); Study Completion 2018-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norman Brest, MD, Principal Investigator
Locations (1):
- Lankenau Medical Center, Wynnewood, Pennsylvania, United States

REFERENCES:
- [Background] Nelson G, Kalogera E, Dowdy SC. Enhanced recovery pathways in gynecologic oncology. Gynecol Oncol. 2014 Dec;135(3):586-94. doi: 10.1016/j.ygyno.2014.10.006. Epub 2014 Oct 12. PMID 25316179
- [Background] Moore A, Costello J, Wieczorek P, Shah V, Taddio A, Carvalho JC. Gabapentin improves postcesarean delivery pain management: a randomized, placebo-controlled trial. Anesth Analg. 2011 Jan;112(1):167-73. doi: 10.1213/ANE.0b013e3181fdf5ee. Epub 2010 Nov 16. PMID 21081764
- [Background] Dowell D, Haegerich TM, Chou R. CDC Guideline for Prescribing Opioids for Chronic Pain--United States, 2016. JAMA. 2016 Apr 19;315(15):1624-45. doi: 10.1001/jama.2016.1464. PMID 26977696
- [Background] Committee opinion no. 633: Alcohol abuse and other substance use disorders: ethical issues in obstetric and gynecologic practice. Obstet Gynecol. 2015 Jun;125(6):1529-1537. doi: 10.1097/01.AOG.0000466371.86393.9b. PMID 26000541
- [Background] Sachs HC; Committee On Drugs. The transfer of drugs and therapeutics into human breast milk: an update on selected topics. Pediatrics. 2013 Sep;132(3):e796-809. doi: 10.1542/peds.2013-1985. Epub 2013 Aug 26. PMID 23979084
- [Background] Wheeler M, Oderda GM, Ashburn MA, Lipman AG. Adverse events associated with postoperative opioid analgesia: a systematic review. J Pain. 2002 Jun;3(3):159-80. doi: 10.1054/jpai.2002.123652. No abstract available. PMID 14622770
- [Background] Guttuso T Jr, Shaman M, Thornburg LL. Potential maternal symptomatic benefit of gabapentin and review of its safety in pregnancy. Eur J Obstet Gynecol Reprod Biol. 2014 Oct;181:280-3. doi: 10.1016/j.ejogrb.2014.08.013. Epub 2014 Aug 17. PMID 25195202
- See also: Related Info — http://erassociety.org/
- See also: Related Info — https://www.cdc.gov/nchs/fastats/delivery.htm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Alternate Management | Control
Started ("Reason Not Completed" was reported in aggregate - this data was not recorded as separate rows per reason.) | 641 | 853
Completed | 475 | 571
Not Completed | 166 | 282
Not completed — Received general anesthesia, Explarel or Naloxone; Return to OR; switched groups | 166 | 282

BASELINE CHARACTERISTICS:
Population: Baseline Measures were only recorded and analyzed for the participants who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Alternate Management | Control | Total
Number analyzed (Participants) | 475 | 571 | 1046
Age, Categorical [Count of Participants; unit: Participants] — Baseline Measures were only recorded and analyzed for the participants who completed the study
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 475 | 571 | 1046
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Baseline Measures were only recorded and analyzed for the participants who completed the study
  years | 32.4 (5.0) | 31.9 (4.7) | 32.1 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline Measures were only recorded and analyzed for the participants who completed the study
  Participants
    Female | 475 | 571 | 1046
    Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Baseline Measures were only recorded and analyzed for the participants who completed the study Population: Baseline Measures were only recorded and analyzed for the participants who completed the study
  Participants
    American Indian or Alaska Native | 4 | 3 | 7
    Asian | 14 | 34 | 48
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 142 | 141 | 283
    White | 302 | 370 | 672
    More than one race | 3 | 10 | 13
    Unknown or Not Reported | 10 | 13 | 23
Region of Enrollment [Number; unit: participants]
  United States | 475 | 571 | 1046

OUTCOME MEASURES:

1. Primary Outcome: Narcotic Utilization
Description: total narcotic utilization measured with Morphine Milligram Equivalent (MME)
  The conversion scale being used will be the Center for Disease Control and Prevention Morphine Equivalent Score.
  Lower scores represent less opioid use and a better outcome. Higher scores represent more opioid use and a worse outcome.
Time Frame: From time of consent until hospital discharge (3 days)
Measure: Mean (Standard Deviation); unit: MME
Arm/Group | Alternate Management | Control
Number analyzed (Participants) | 476 | 641
MME | 33.3 (52.4) | 47.2 (60.4)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded, per patient, from time of consent until hospital discharge (3 days)
Arm/Group | Alternate Management | Control
All-Cause Mortality (participants affected / at risk) | 0/475 | 0/641
Serious Adverse Events (participants affected / at risk) | 0/475 | 0/641
Other Adverse Events (participants affected / at risk) | 0/475 | 0/641

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-30): https://cdn.clinicaltrials.gov/large-docs/19/NCT03330119/Prot_SAP_001.pdf